CLINICAL TRIAL: NCT04141098
Title: Lumbar Operatively Inserted PerQdisc Artificial Implant Following Nuclectomy - LOPAIN1
Brief Title: Lumbar Operatively Inserted PerQdisc Artificial Implant Following Nuclectomy
Acronym: LOPAIN1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical trial was terminated prematurely due to receipt of CE mark
Sponsor: Spinal Stabilization Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-003
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Disc Disease; Chronic Low-back Pain
Keywords: Degenerative Disc Disease; DDD; Chronic Low-back Pain; Disc Herniation; Nucleus Replacement; Low back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is an open-label study. Patients will receive one implant if they meet all inclusion/exclusion criteria after a review by the Medical Advisory Board (MAB). Patients that cannot receive the implant due to an intraoperative exclusion, will receive standard of care treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Total Nucleus Replacement (Experimental): All patients that meet the inclusion/exclusion criteria will receive the PerQdisc® Nucleus Replacement Device.
  Interventions: Device: All patients that meet the inclusion/exclusion criteria will receive the PerQdisc® Nucleus Replacement Device.

INTERVENTIONS:
Device: All patients that meet the inclusion/exclusion criteria will receive the PerQdisc® Nucleus Replacement Device. — All patients meeting all inclusion criteria and no exclusion criteria will be considered for nucleus replacement surgery following a review by the Medical Advisory Board. Any patient meeting any of the three intraoperative exclusion criteria will receive an alternative standard of care therapy.

SUMMARY:
This study will be a prospective, open-label, multi-center study that will collect safety data for the minimally invasive PerQdisc Nucleus Replacement Device deployed to reduce chronic low back pain.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, multi-center study that will collect safety and efficacy data for the minimally invasive PerQdisc Nucleus Replacement Device (NRD). Patients will have degenerative disc disease (DDD) in one or more lumbar discs. The NRD is used for surgical replacement of a single nucleus pulposus between spinal lumbar discs L1-S1 using an anterior or lateral transpsoas approach. Currently the surgical gold standard involves spinal fusion of the affected vertebral bodies, reducing range of motion and increasing stress on other vertebral bodies. The goal of nucleus replacement is to reduce chronic low back pain by maintaining disc height while preserving range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature and between 21 and 60 years of age.
* Patient has Degenerative Disc Disease (DDD) at one or more levels between L1 and S1
* History and clinical findings suggestive of symptomatic DDD:

Darkened disc on MRI in T2 weighted images Patients with at least 6 months of low back pain (location defined as the space between the lower margin of the posterior rib cage and horizontal gluteal fold) that is resistant to nonsurgical conservative therapy.

* Patient has adequate disc height (~6mm) at the level to be treated
* Patient has pre-operative Oswestry Low Back Disability score of greater than or equal to 40 (0-100 scale).
* Patient has pre-operative back pain VAS score of greater than or equal to 40 (0-100 scale)
* Patient has received conservative, non-surgical treatment for back pain for a minimum of 6 months.
* Patient has signed the approved Informed Consent Form.

Exclusion Criteria:

* Patient has had prior lumbar spine surgery
* Spinal fusion at any level
* Patient has ankylosing spondylitis or other spondyloarthropathy.
* Patient has isthmic spondylolisthesis or degenerative spondylolisthesis greater than 2 mm.
* Patient has congenital moderate or severe spinal stenosis or epidural lipomatosis.
* Patient has significant facet disease.
* Patient has had prior lumbar spine surgery
* Spinal fusion at any level
* Patient has any known active malignancy.
* Patient has previously undergone or currently on immunosuppressive therapy. Steroids used to treat inflammation are allowed.
* Patient has active local or systemic infection.
* Patient has been diagnosed with hepatitis, rheumatoid arthritis, lupus erythematosus, or other autoimmune disease, including AIDS, ARC and HIV.
* Patient has diabetes mellitus (Type 1 or 2), requiring daily insulin management.
* Patient is pregnant or plans to become pregnant during the course of the study. Pregnancy ruled out by urine or serum HCG.
* Patient has a known allergy to silicone (polymer and balloon material) or barium sulfate (polymer).
* Patient participated in another investigational drug or device study within the past 30 days.
* Patient belongs to a vulnerable population or has a condition such that his/her ability to provide informed consent, comply with follow-up requirements, or provide self- assessments is compromised (e.g. developmentally disabled, prisoner, chronic alcohol/ substance abuser)
* Patient has a significant disc herniation at the level to be treated
* Patient has a significant Schmorl's node in the level to be treated

Intraoperative exclusion criteria:

* Protrusion of the 20A imaging balloon up to or beyond the outer margin of the vertebra during the imaging steps.
* Patient has a violated endplate as determined by imaging balloon during fluoroscopy
* Patient has a disc space that is too narrow for implantation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Post surgical change in degree of disability | 6 months
  Patient reported outcomes for degree of disability will be monitored using the Oswestry Disability Index (scale of 0-100). Higher scores indicate greater level of disability.
Post surgical change in back pain: Visual Analogue Scale | 6 months
  Patient reported outcomes will be reported using the Visual Analogue Scale (0-100mm). Higher scores indicate greater levels of back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hess, MD, Study Chair — London Spine Clinic/ATOS-Klinik; Jeff Golan, MD, Study Chair — Jewish General Hospital
Locations (1):
- Sanatorio Americano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No